CLINICAL TRIAL: NCT06647004
Title: Relationship of Dorsal Flexion, Static Balance and Isometric Strength of Abductors and Adductors in Inline Skaters. Observational Study.
Brief Title: Inline Skaters Observational Study.
Status: Completed | Type: Observational
Sponsor: Javier Reina Abellan; PhD (Other)
Responsible Party: Sponsor-Investigator, Javier Reina Abellan; PhD, Doctor in Teaching and Educational Innovation, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Other Study IDs: TESIS LARA
Record Dates: First submitted 2024-10-08; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Range of Motion, Articular; Strength; Balance
Keywords: Inline Skaters; Static Balance; Strength; Dorsiflexion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inline Skaters: Amateur In-line skaters aged between 18 and 59 years, with at least one year of experience, without serious illnesses in the last six months or pharmacological treatments that could alter sports practice.

SUMMARY:
The study analyzes the relationship of ankle dorsiflexion, static balance and maximum isometric strength of abductors and adductors in amateur inline skaters, and then make a comparison between sexes.

DETAILED DESCRIPTION:
Inline skating has grown fastly and been adopted as a new form of exercise. Its relative novelty has led to research focusing on associated injuries and protective measures. The synthesis of information carried out on studies about other modalities of skating has allowed us to highlight the physical skills necessaries because of the high demand of its practice; as well as the strength in the lower limbs and the ability to balance, abilities related to each other and associated with better performance of the athlete. The use of the skating boot has also been the subject of study due to the mobility limitations that its rigidity could cause and the repercussions that such deficits would have on the injuries and abilities of skaters.

The main objective of this research will be to analyze the relationship between ankle dorsiflexion mobility, static balance and abductor and adductor strength in skaters. As well as compare the data obtained between both sexes.

The subjects who will make up the sample will be intermediate level amateur inline skaters, of both sexes and aged between 18 and 59 years; with at least one year of experience and who skate with a frequency equal to or greater than three days per week. Ankle dorsiflexion mobility, static balance and maximum isometric strength of abductors and adductors will be analyzed. The data obtained will be studied to assess the possible relationship between the abilities examined. Finally, a comparison between sexes will be made.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 59 years.
* Minimum one year of experience.
* Sports practice at least 1 day a week.

Exclusion Criteria:

* Surgical interventions in the lower limbs during the 6 months prior to the study.
* Illness or ingestion of drugs that may alter sports practice.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Amateur Inline Skaters of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Ankle Dorsiflexion | A single measurement was conducted prior to one of the weekly practices and at least 24 hours after the last practice between May and September, during the months in which data collection took place.
  Test to assess ankle dorsiflexion, performing 3 attempts and keeping the best result. The Gyko (Microgate S.r.I, Italy) device was positioned on the tibia about ten centimeters below the knee of the dominant leg. All of them had to perform a squat with their upper limbs extended above their heads and without taking their heels off the ground. The speed of execution was that preferred by each subject.
Static Balance | A single measurement was conducted prior to one of the weekly practices and at least 24 hours after the last practice between May and September, during the months in which data collection took place.
  To evaluate static balance, three fifteen-second measurements were made on the dominant leg. With thirty seconds of rest on both feet in between. Then the final result was calculated based on the data collected from each repetition by Footscan® V9 Software. During the test, the patient was asked to position himself on the Footscan® Pressure Platform (without shoes or socks), so that the second toe of the supporting leg was aligned with the antero-posterior line of the platform, and the medial malleolus with the latero-medial line. The opposite leg, suspended in the air, must maintain a 90º knee bend and the arms must remain crossed over the chest.
  First, the static balance assessment was completed with eyes open, during which participants were asked to look at a fixed point, located approximately five meters away. Then the evaluation proceeded with eyes closed, following the same steps.
Isometric Maximum Strength | A single measurement was conducted prior to one of the weekly practices and at least 24 hours after the last practice between May and September, during the months in which data collection took place.
  The maximum isometric strength of adductors and abductors of the dominant leg of each participant, in the supine position on a medical stretcher. Subjects were instructed to grab both sides of the stretcher to stabilize themselves. Accessory movements were not allowed with any part of the body during the test.
  After receiving the instructions, they were asked to perform a maximum isometric contraction of five seconds against the dynameter (Nicholas Manual Muscle Tester, Lafayette Indiana Instruments) with the belt hugging their lower limb five centimeters away from the lateral and medial malleolus to measure abduction and adduction, respectively. The participants were guided by the hand of the researchers to ensure that the correct action was taken. In addition, verbal stimuli were used to encourage the subjects. The dynamometer was fixed by a belt to a stable and vertical structure anchored to the ground.

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Sánchez Torres, Torre del Mar, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No